CLINICAL TRIAL: NCT04636086
Title: Vitamin D Supplementation and Covid-19: a Randomised, Double- Blind, Controlled Study
Brief Title: Effect of Vitamin D on Hospitalized Adults With COVID-19 Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Liege (Other)
Collaborators: Laboratoires SMB S.A. (Industry)
Responsible Party: Principal Investigator, Anne-Françoise Rousseau, Head of Clinic, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D-COVID
Record Dates: First submitted 2020-11-17; First posted 2020-11-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test treatment (Experimental): Test Treatment: Ampoule for enteral use containing 25,000 IU/mL of cholecalciferol taken according to the following scheme: one ampoule on Day 1, Day 2, Day 3, Day 4, Day 8, Day 15, Day 22, Day 29 and Day 36.
  Interventions: Drug: Cholecalciferol
- Placebo treatment (Placebo Comparator): Placebo Treatment: Ampoule of placebo for enteral use containing excipient only taken according to the following scheme: one ampoule on Day 1, Day 2, Day 3, Day 4, Day 8, Day 15, Day 22, Day 29 and Day 36.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Cholecalciferol — Vitamin D supplementation
  Other Names: D-Cure
  Arms: Test treatment
Other: Placebo — Placebo comparator
  Arms: Placebo treatment

SUMMARY:
The objective of the study is to evaluate the clinical efficacy and safety of vitamin D supplementation in hospitalized patients with COVID-19.

DETAILED DESCRIPTION:
Phase IV, interventional, randomised, double blind, placebo-controlled and parallel study to evaluate the clinical efficacy and safety of vitamin D supplementation in hospitalized patients with COVID-19.

Patients will participate in the study for a maximum of 9 weeks, which includes an up to 6-week treatment period and a maximum of 3-week follow-up period.

A total of 100 (50 in each group) patients will be randomized in the study and will either receive the test treatment or the placebo treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female over 18 years old (18 years inclusive).
* Has laboratory-confirmed SARS-CoV-2 infection as determined by PCR, or other commercial or public health assay in any specimen as diagnosed within 72 hours prior to randomization.
* Expected to survive for at least 96 hours after study entry.
* If patient is a female of childbearing potential, patient must use an effective means of birth control (oral, intravaginal or transdermal oestrogen-progestogen combined hormonal contraceptives or intrauterine devices or sexual abstinence).
* Subject or legally authorized representative understands and agrees to comply with planned study procedures.
* Subject or legally authorized representative provides informed consent prior to initiation of any study procedures.

Exclusion Criteria:

* Women currently pregnant or breast-feeding.
* Patients presenting acute impairment of renal function or nephrolithiasis.
* Patients presenting hypercalcaemia and/or hypercalciuria
* Patients presenting pseudohypoparathyroidism
* Use of any vitamin D supplementation alone or in association at screening visit;
* Use of any prohibited medication as detailed in the concomitant medication section
* Patients with any sensitivity or allergy to any of the products used within this clinical trial.
* Presence of any other condition or illness, which, in the opinion of the investigator, would interfere with optimal participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2022-04-10 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Vitamin D serum concentration | Baseline, on days 8, 15, 22, 29 (+/-1 day), or last day of hospitalization, and finally at day 15 to 30 after hospital discharge
  Mean change from screening to end of treatment phase in 25(OH)D3 serum concentration

SECONDARY OUTCOMES:
Clinical improvement | Baseline and up to 4 weeks after randomization on days 8, 15, 22, 29 (+/-1 day), or last day of hospitalization, and finally at day 15 to 30 after hospital discharge
  Ordinal scale for clinical improvement as recommended by WHO
Hospital length of stay. | at day 15 to 30 after hospital discharge
  Hospital length of stay.
Intensive care unit length of stay. | at day 15 to 30 after hospital discharge
  Intensive care unit length of stay.
Supplemental oxygen, non-invasive or invasive ventilation or organ support | Baseline and up to 4 weeks after randomization on days 8, 15, 22, 29 (+/-1 day), or last day of hospitalization, and finally at day 15 to 30 after hospital discharge
  Number of patients requiring supplemental oxygen, non-invasive ventilation or high flow oxygen devices, invasive mechanical ventilation or additional organ support (pressors, renal replacement therapy, extracorporeal membrane oxygenation).
Duration of supplemental oxygen, non-invasive or invasive ventilation or organ support | at day 15 to 30 after hospital discharge
  Duration of any organ support
Absence of fever | Last day of hospitalization, or at at day 15 to 30 after hospital discharge
  Time until absence of fever for more than 48h without antipyretics.
Time until negative laboratory SARS-CoV-2 test. | Last day of hospitalization , or at at day 15 to 30 after hospital discharge
  Time until negative laboratory SARS-CoV-2 test.
Mortality all causes. | Last day of hospitalization , or at at day 15 to 30 after hospital discharge
  Mortality all causes.
Mortality related to Covid-19. | Last day of hospitalization , or at at day 15 to 30 after hospital discharge
  Mortality related to Covid-19.
Biological markers | Baseline, on days 8, 15, 22, 29 (+/-1 day), or last day of hospitalization, and finally at day 15 to 30 after hospital discharge
  Blood levels of C-reactive protein, interleukin 6 and 10, cathelicidin, white blood cells, creatinin and 1,25(OH)2-D3

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amrein K, Zajic P, Schnedl C, Waltensdorfer A, Fruhwald S, Holl A, Purkart T, Wunsch G, Valentin T, Grisold A, Stojakovic T, Amrein S, Pieber TR, Dobnig H. Vitamin D status and its association with season, hospital and sepsis mortality in critical illness. Crit Care. 2014 Mar 24;18(2):R47. doi: 10.1186/cc13790. PMID 24661739
- [Background] Amrein K, Litonjua AA, Moromizato T, Quraishi SA, Gibbons FK, Pieber TR, Camargo CA Jr, Giovannucci E, Christopher KB. Increases in pre-hospitalization serum 25(OH)D concentrations are associated with improved 30-day mortality after hospital admission: A cohort study. Clin Nutr. 2016 Apr;35(2):514-521. doi: 10.1016/j.clnu.2015.03.020. Epub 2015 Apr 14. PMID 25935851
- [Background] Amrein K, Schnedl C, Holl A, Riedl R, Christopher KB, Pachler C, Urbanic Purkart T, Waltensdorfer A, Munch A, Warnkross H, Stojakovic T, Bisping E, Toller W, Smolle KH, Berghold A, Pieber TR, Dobnig H. Effect of high-dose vitamin D3 on hospital length of stay in critically ill patients with vitamin D deficiency: the VITdAL-ICU randomized clinical trial. JAMA. 2014 Oct 15;312(15):1520-30. doi: 10.1001/jama.2014.13204. PMID 25268295
- [Background] Barlow PG, Beaumont PE, Cosseau C, Mackellar A, Wilkinson TS, Hancock RE, Haslett C, Govan JR, Simpson AJ, Davidson DJ. The human cathelicidin LL-37 preferentially promotes apoptosis of infected airway epithelium. Am J Respir Cell Mol Biol. 2010 Dec;43(6):692-702. doi: 10.1165/rcmb.2009-0250OC. Epub 2010 Jan 22. PMID 20097832
- [Background] Barnett N, Zhao Z, Koyama T, Janz DR, Wang CY, May AK, Bernard GR, Ware LB. Vitamin D deficiency and risk of acute lung injury in severe sepsis and severe trauma: a case-control study. Ann Intensive Care. 2014 Feb 24;4(1):5. doi: 10.1186/2110-5820-4-5. PMID 24559079
- [Background] Beard JA, Bearden A, Striker R. Vitamin D and the anti-viral state. J Clin Virol. 2011 Mar;50(3):194-200. doi: 10.1016/j.jcv.2010.12.006. Epub 2011 Jan 15. PMID 21242105
- [Background] Braun AB, Gibbons FK, Litonjua AA, Giovannucci E, Christopher KB. Low serum 25-hydroxyvitamin D at critical care initiation is associated with increased mortality. Crit Care Med. 2012 Jan;40(1):63-72. doi: 10.1097/CCM.0b013e31822d74f3. PMID 21926604
- [Background] Cavalier E, Fache W, Souberbielle JC. A Randomised, Double-Blinded, Placebo-Controlled, Parallel Study of Vitamin D3 Supplementation with Different Schemes Based on Multiples of 25,000 IU Doses. Int J Endocrinol. 2013;2013:327265. doi: 10.1155/2013/327265. Epub 2013 Jan 28. PMID 23431293
- [Background] Abhimanyu, Coussens AK. The role of UV radiation and vitamin D in the seasonality and outcomes of infectious disease. Photochem Photobiol Sci. 2017 Mar 16;16(3):314-338. doi: 10.1039/c6pp00355a. PMID 28078341
- [Background] Dancer RC, Parekh D, Lax S, D'Souza V, Zheng S, Bassford CR, Park D, Bartis DG, Mahida R, Turner AM, Sapey E, Wei W, Naidu B, Stewart PM, Fraser WD, Christopher KB, Cooper MS, Gao F, Sansom DM, Martineau AR, Perkins GD, Thickett DR. Vitamin D deficiency contributes directly to the acute respiratory distress syndrome (ARDS). Thorax. 2015 Jul;70(7):617-24. doi: 10.1136/thoraxjnl-2014-206680. Epub 2015 Apr 22. PMID 25903964
- [Background] Guo YR, Cao QD, Hong ZS, Tan YY, Chen SD, Jin HJ, Tan KS, Wang DY, Yan Y. The origin, transmission and clinical therapies on coronavirus disease 2019 (COVID-19) outbreak - an update on the status. Mil Med Res. 2020 Mar 13;7(1):11. doi: 10.1186/s40779-020-00240-0. PMID 32169119
- [Background] De Niet S, Coffiner M, Da Silva S, Jandrain B, Souberbielle JC, Cavalier E. A Randomized Study to Compare a Monthly to a Daily Administration of Vitamin D(3) Supplementation. Nutrients. 2018 May 23;10(6):659. doi: 10.3390/nu10060659. PMID 29882841
- [Background] Gombart AF, Pierre A, Maggini S. A Review of Micronutrients and the Immune System-Working in Harmony to Reduce the Risk of Infection. Nutrients. 2020 Jan 16;12(1):236. doi: 10.3390/nu12010236. PMID 31963293
- [Background] Grant WB, Lahore H, McDonnell SL, Baggerly CA, French CB, Aliano JL, Bhattoa HP. Evidence that Vitamin D Supplementation Could Reduce Risk of Influenza and COVID-19 Infections and Deaths. Nutrients. 2020 Apr 2;12(4):988. doi: 10.3390/nu12040988. PMID 32252338
- [Background] Greiller CL, Martineau AR. Modulation of the immune response to respiratory viruses by vitamin D. Nutrients. 2015 May 29;7(6):4240-70. doi: 10.3390/nu7064240. PMID 26035247
- [Background] Gruber-Bzura BM. Vitamin D and Influenza-Prevention or Therapy? Int J Mol Sci. 2018 Aug 16;19(8):2419. doi: 10.3390/ijms19082419. PMID 30115864
- [Background] Han JE, Jones JL, Tangpricha V, Brown MA, Brown LAS, Hao L, Hebbar G, Lee MJ, Liu S, Ziegler TR, Martin GS. High Dose Vitamin D Administration in Ventilated Intensive Care Unit Patients: A Pilot Double Blind Randomized Controlled Trial. J Clin Transl Endocrinol. 2016 Jun;4:59-65. doi: 10.1016/j.jcte.2016.04.004. Epub 2016 May 5. PMID 27419080
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Yim S, Dhawan P, Ragunath C, Christakos S, Diamond G. Induction of cathelicidin in normal and CF bronchial epithelial cells by 1,25-dihydroxyvitamin D(3). J Cyst Fibros. 2007 Nov 30;6(6):403-10. doi: 10.1016/j.jcf.2007.03.003. Epub 2007 Apr 27. PMID 17467345
- [Derived] Shakoor H, Feehan J, Al Dhaheri AS, Cheikh Ismail L, Ali HI, Alhebshi SH, Apostolopoulos V, Stojanovska L. Role of vitamin D supplementation in aging patients with COVID-19. Maturitas. 2021 Oct;152:63-65. doi: 10.1016/j.maturitas.2021.03.006. Epub 2021 Mar 16. No abstract available. PMID 33757717